CLINICAL TRIAL: NCT01564888
Title: Prevention of Radial Artery Occlusion: Prophylactic Hyperperfusion Evaluation Trial
Acronym: PROPHET-II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Total Cardiovascular Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MIL/IMRC/TCC/TP/10/2010
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Occlusion of Artery
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patent hemostasis (Placebo Comparator): Patent hemostasis is the technique for radial artery hemostasis after transradial catheterization, with proactive attempt to maintain radial artery hemostasis and radial artery patency.
  Interventions: Procedure: Ulnar artery compression
- Ulnar artery compression (Active Comparator): Ulnar artery compression will involve radial artery hemostasis using patent hemostasis technique and compression of ulnar artery to the point of occluding flow, in an attempt to augment radial artery flow.
  Interventions: Procedure: Ulnar artery compression

INTERVENTIONS:
Procedure: Ulnar artery compression — Compression of ulnar artery for 2 hours with radial artery hemostasis

SUMMARY:
Evaluating the effect of ulnar artery compression while pressing on radial artery to stop bleeding, in maintaining radial artery potency, after cardiac catheterization through the radial artery. We prospectively plan to compare 3000 patients referred for cardiac catheterization, randomized into two groups, one group receiving radial artery compression for stopping bleeding, in a standard fashion following best practices, and the other group receiving radial artery compression using standard best practices and ulnar artery compression. Radial artery status will be evaluated in 24 hours and 30 days of the procedure to evaluate its potency, using plethysmography.

ELIGIBILITY:
Inclusion Criteria:

* patients referred for diagnostic cardiac catheterization.

Exclusion Criteria:

* previous ipsilateral radial artery puncture, warfarin therapy, absence of intact palmar collateral circulation, scleroderma, ipsilateral radial artery surgery, lone upper extremity (contralateral upper extremity amputation), ipsilateral upper extremity chronic pain.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2011-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
30 day radial artery occlusion | 30 days
  Evaluation of radial artery patency using plethysmography

SECONDARY OUTCOMES:
hand ischemia | 2 hours
  evaluated by clinical evaluation for neurosensory deficit or other clinical signs of ischemia.

CONTACTS AND LOCATIONS:
Overall Officials: Samir B Pancholy, MD, Principal Investigator
Locations (2):
- University Hospital and Faculty of Medicine, Pilsen, Czechia
- V.S. General hospital, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No